CLINICAL TRIAL: NCT07092709
Title: Tenecteplase for Intravenous Stroke Thrombolysis in Recent DOAC Users (PEARL-DOAC): A Multicenter, Prospective, Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Tenecteplase for Intravenous Stroke Thrombolysis in Recent DOAC Users
Acronym: PEARL-DOAC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSKY-2025-484-01
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous tenecteplase (Experimental)
  Interventions: Drug: Tenecteplase (TNK) (0.25 mg/kg, to maximum of 25mg)
- Matched placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenecteplase (TNK) (0.25 mg/kg, to maximum of 25mg) — Tenecteplase is administered as a single intravenous bolus at a dose of 0.25 mg/kg, with a maximum of 25 mg, administered as soon as possible after the randomization, and within 24 hours of stroke onset.
  Arms: Intravenous tenecteplase
Drug: Placebo — Matched placebo is administered as a single intravenous bolus at a dose of 0.25 mg/kg, with a maximum of 25 mg, administered as soon as possible after the randomization, and within 24 hours of stroke onset.
  Arms: Matched placebo

SUMMARY:
An investigator-initiated, multicenter, randomized, placebo-controlled, double-blind trial to determine the efficacy and safety of intravenous tenecteplase thrombolysis in acute ischemic stroke (AIS) patients with recent direct oral anticoagulants (DOACs) intake in improving the 90-day functional outcome.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized, double-blind, placebo-controlled clinical trial designed to evaluate the efficacy and safety of intravenous tenecteplase thrombolysis in AIS patients with recent DOACs intake 48 hours prior to enrollment. The primary outcome is the proportion of patients with a 90-day modified Rankin scale (mRS) of 0-1.

Study intervention: (1) Participants in the intervention group will receive tenecteplase administered as a single intravenous bolus at a dose of 0.25 mg/kg, with a maximum of 25 mg, administered as soon as possible after the randomization. (2) Participants in the control group will receive matched intravenous placebo in the same approach. All participants will receive standard medical treatment.

A total of 912 participants are anticipated to be recruited for this study, with 456 participants in each group (1:1 ratio).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Clinically diagnosed with acute ischemic stroke.
3. DOACs intake within 48 hours prior to enrollment, or on an ongoing DOACs therapy but the exact time of last intake is unknown.

   * To ensure a representative study population, the investigators will limit the number of patients who took DOACs within 24-48 hours before enrollment or those with unknown last intake time to 50% of the planned sample size. If this number is reached, the inclusion criterion 3 will be modified:

   DOACs intake within 24 hours prior to enrollment.
4. Study intervention (IVT or placebo) can be started

   1. within 4.5 hours of last known well (LKW). OR
   2. within 4.5 to 24 hours of LKW (including wake-up stroke) AND evidence of target mismatch profile on CT perfusion or MR perfusion (ischemic core volume < 50mL, hypoperfused volume to ischemic core volume ratio > 1.6, mismatch volume ≥10ml).

      * Hypoperfused tissue is defined as Tmax >6s on CT perfusion or MR perfusion. Ischemic core is defined as rCBF <30% on CT perfusion or ADC<620μm^2/s on diffusion MRI.
5. Baseline National Institutes of Health Stroke Scale (NIHSS) 4-25. OR Disabling stroke with baseline NIHSS of 0-3, including complete hemianopia, aphasia, measurable deficit on motor power, or other disabling neurological deficit judged by the investigator.
6. Written informed consent signed by patients or their legally authorized representatives.

Exclusion Criteria:

1. Intracranial or subarachnoid hemorrhage confirmed by cranial computed tomography (CT) or magnetic resonance imaging (MRI), or any intracranial hemorrhage history.
2. Allergic to tenecteplase.
3. Pre-stroke mRS≥2
4. Planned endovascular treatment.
5. Currently on dual antiplatelet therapy in addition to DOAC therapy.
6. Planned DOAC reversal treatment (including Idarucizumab, Andexanet and tranexamic acid).
7. Hypodensity on non-contrast CT estimates to be ≥ 1/3 MCA territory.
8. Severe head trauma or other severe trauma in the last 3 months.
9. Intracranial tumor, arteriovenous malformation and large-size aneurysm (≥10 mm) found before enrollment.
10. Intracranial surgery, intraspinal surgery or other major surgeries within 3 months before enrollment (based on the assessment of the investigators)
11. Gastrointestinal or urinary system hemorrhage within the past 3 weeks.
12. Active visceral bleeding.
13. Aortic arch dissection confirmed by examination or medical history.
14. Infective endocarditis confirmed by examination or medical history.
15. Platelet count less than 100 × 10^9 /L.
16. Patients received heparin or low-molecular-weighted heparin treatment within 24h before enrollment.
17. Pregnant or lactating women.
18. Blood glucose <50 mg/dl (2.78mmol/L) or >400 mg/dl (22.2mmol/L) during screening.
19. Uncontrolled hypertension with persistent systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg, refractory to medical management.
20. Life expectancy less than 6 months due to malignancy, severe cardiopulmonary disease, or other terminal illness.
21. Participating in other trials.
22. Other conditions deemed unsuitable for the study by the investigator, such as inability to comprehend or comply with study procedures or follow-up due to mental illness, cognitive or emotional disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The modified Rankin Scale score (mRS) 0-1 | 90 (±14) days
  The proportion of mRS score 0-1 at 90 (±14) days.

SECONDARY OUTCOMES:
The modified Rankin Scale score (mRS) 0-2 | 90 (±14) days
  The proportion of mRS score 0-2 at 90 (±14) days.
The modified Rankin Scale score (mRS) 0-3 | 90 (±14) days
  The proportion of mRS score 0-3 at 90 (±14) days
Level of disability | 90 (±14) days
  The shift analysis of the 90-day mRS with 5-6 merged at 90 (±14) days.
The proportion of NIHSS 0-1 or ≥4 points reduction | 24 (±12) hours
  The proportion of NIHSS 0-1 or ≥4 points reduction at 24 (±12) hours.
Quality of life (EQ-5D-5L) | 90 (±14) days
  Quality of life measured by EQ-5D-5L scale score at 90 (±14) days.
Neurologic deficit (NIHSS score) changes | 7 (±1) days or at discharge
  Neurologic deficit (NIHSS score) changes from baseline to 7 (±1) days or at discharge if earlier.

OTHER OUTCOMES:
SAFETY OUTCOME: Symptomatic intracranial hemorrhage | 24 (±12) hours
  Rate of symptomatic intracranial hemorrhage (sICH) within 36 hours from randomization (European Cooperative Acute Stroke Study [ECASS] III classification)
SAFETY OUTCOME: Any intracranial hemorrhage | 24 (±12) hours
  Rate of any intracranial hemorrhage within 36 hours from randomization (ECASS-III classification)
SAFETY OUTCOME: Major extracranial bleeding | 24 (±12) hours
  Rate of major extracranial bleeding within 36 hours from randomization (as defined by the Global Utilization of Streptokinase and Tissue-type Plasminogen Activator for Occluded Coronary Arteries, GUSTO criteria: moderate and severe bleeding)
SAFETY OUTCOME: Mortality | 90(±14) days
  All-cause mortality within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Raul G. Nogueira, Principal Investigator — UPMC Stroke Institute, Departments of Neurology and Neurosurgery, University of Pittsburgh
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available from Principal Investigators (Prof. Yamei Tang and Prof. Raul G. Nogueira) upon reasonable request 6 months after the trial completion.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the trial completion.
Access Criteria: The IPD will be available from Principal Investigators (Prof. Yamei Tang and Prof. Raul G. Nogueira) upon reasonable request.